CLINICAL TRIAL: NCT01002586
Title: Wii-Fit For Improving Activity, Gait And Balance In Alzheimer's Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0361-09-EP
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer's Dementia; Falls; Gait Impairment; Balance Impairment
Keywords: Alzheimer's dementia; Wii-Fit; Walking; Falls
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wii-Fit arm (Experimental): Half hour daily, five days a week, for 8 weeks
  Interventions: Other: Wii-Fit intervention
- Walking arm (Active Comparator): Half hour daily, five days a week, for 8 weeks
  Interventions: Other: Walking exercise program

INTERVENTIONS:
Other: Wii-Fit intervention — Half hour daily, five days a week, for 8 weeks
  Other Names: Exercise intervention
  Arms: Wii-Fit arm
Other: Walking exercise program — walking exercise program
  Arms: Walking arm

SUMMARY:
Alzheimer's Dementia (AD) contributes to poor balance, impaired gait and functional status, thereby, increasing the risk of falls. AD is an independent risk factor for hip fractures. Those with balance problems and gait impairments are at higher risk for long term placement and death related to falls. Exercise interventions improve gait and balance in the elderly. In participants with existing AD, physical activity has shown to prevent further cognitive decline and improve quality of life and prevent falls. However, it is difficult to engage patients with AD in long term exercise programs. The expense of physical therapy limits its easy accessibility. Use of everyday technology might bridge this gap by providing high level of engagement via the use of multimedia while providing a cost-effective alternative. Wii Fit is one such multimedia platform.

Wii fit is a Nintendo gaming console used for aerobics, strength training and balance activities. This device includes a balance board that senses weight and shifts in movement and balance. Virtual trainers talk the user through the activity while tracking the user's progress. The investigators propose an 8-week prospective randomized study with the treatment group receiving the exercise program delivered by Wii-Fit system and the comparison arm receiving a walking exercise program in a community dwelling setting. Subjects in each arm will participate for 30 minutes daily five days a week.

DETAILED DESCRIPTION:
Alzheimer's Dementia (AD) contributes to poor balance, impaired gait and functional status, thereby, increasing the risk of falls. AD is an independent risk factor for hip fractures. Those with balance problems and gait impairments are at higher risk for long term placement and death related to falls. Gait impairments in those with dementia include shortened step length, increased double support time, step to step variability, and decreased gait speed. These gait impairments worsen with dual tasking probably due to common brain areas involved in gait and other cognitive tasks.

Exercise interventions improve gait and balance in the elderly. In subjects with existing AD, physical activity has shown to prevent further cognitive decline and improve quality of life and prevent falls. However, it is difficult to engage patients with AD in long term exercise programs. The expense of physical therapy limits its easy accessibility. Use of everyday technology might bridge this gap by providing high level of engagement via the use of multimedia while providing a cost effective alternative. Wii Fit is one such multimedia platform.

Wii fit is a Nintendo gaming console used for aerobics, strength training and balance activities. This device includes a balance board that senses weight and shifts in movement and balance. Virtual trainers talk the user through the activity while tracking the user's progress.

Although some skilled nursing facilities have started using Wii game system adjunct to routine physical therapy, there have not been any studies. Anecdotal reports note improvement in balance and social benefits using the Wii Fit program. Physical therapists report the ability to customize Wii for each patient. Wii Fit can be successfully used in a cognitively impaired population. A unique feature of this approach is the enjoyment and enthusiasm that many patients derive which is reflected in high levels of engagement.

The invesitgators propose an 8 week prospective randomized study with the treatment group receiving the exercise program delivered by Wii-Fit system and the comparison arm receiving a walking exercise program in a community dwelling setting. Subjects in each arm will participate for 30 minutes daily five days a week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age ≥ 60
* Diagnosis of mild Dementia of Alzheimer's type (MMSE ≥ 18)
* Community dwelling elders, living at home
* History of fall at least once during the year before the study (without serious injury) or a fear of a future fall
* Presence of caregiver(s)
* Presence of television at home

Exclusion Criteria:

* History of myocardial infarction or TIA or stroke in last 6 months
* Presence of serious psychiatric problems that have impact on memory
* Active cancer or new cancer diagnosis in the last year other than skin cancer
* Medical conditions likely to compromise survival, or ability to participate in the exercise program such as severe congestive heart failure, significant musculoskeletal impairments, recent fracture, joint replacements, or severe chronic pain
* Severe visual or auditory impairment or peripheral neuropathy
* Subjects using wheel chair or assistive device for mobility

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2012-07-06 (Actual); Study Completion 2012-07-06 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | 8 weeks and 16 weeks
  The Berg Balance Scale involves 14 mobility tasks, divided into 3 domains: sitting balance, standing balance, and dynamic balance. In the sitting balance, the task is the evaluation of sitting unsupported. Standing balance consist of standing unsupported, standing with eyes closed, standing with feet together, standing on one foot, turning to look behind, grabbing an object from the floor, reaching forward with outstretched arms, and placing one foot in front of the other. In the last domain, the dynamic balance is evaluated with the individual going from sitting to standing, standing to sitting, transferring, turning 360 degrees, placing one foot on a step. Each task is graded on a 5-point ordinal scale that ranges from 0 to 4 for a maximum score of 56. In general, a score of 0 is given when the individual is unable to perform the task, and a
Biomechanical assessment of balance | 8 weeks and 16 weeks
  Biomechanical assessment of balance - center of pressure is assessed while standing on a force platform.
Biomechanical assessment of gait | 8 weeks and 16 weeks
  Biomechanical assessment of gait - reflective markers attached to anatomical landmarks are tracked with motion capture cameras that provide body segment position data as subjects walk on a treadmill. The position data is then used to calculate joint movements, velocities, etc.

SECONDARY OUTCOMES:
Activities of daily living (ADL) | 8 weeks and 16 weeks
  The Activities of Daily Living are a series of basic activities necessary for independent living at home or in the community. They are performed on a daily basis. There are 5 basic categories.
  1. Personal hygiene - bathing/showering, grooming, nail care, and oral care.
  2. Dressing - being able to make appropriate clothing decisions and physically dress and undress oneself.
  3. Eating - the ability to feed oneself, though not necessarily the capability to prepare food.
  4. Maintaining continence - being able to mentally and physically use a restroom. This includes the ability to get on and off the toilet and cleaning oneself.
  5. Transferring/Mobility- being able to stand from a sitting position, as well as get in and out of bed. The ability to walk independently from one location to another.
  These are rated on the basis of the level of independence - a) can be performed independently, b) some assistance needed and c) complete assistance needed.
Instrumental activities of daily living (IADL) | 8 weeks and 16 weeks
  Instrumental Activities of Daily Living are important to being able to live independently, but are not necessarily required on a daily basis. The IADLs include:
  1. Basic communication skills - such as using a regular phone, mobile phone, email, or the internet.
  2. Transportation - either by driving oneself, arranging rides, or the ability to use public transportation.
  3. Meal preparation - meal planning, cooking, clean up, storage, and the ability to safely use kitchen equipment and utensils.
  4. Shopping - the ability to make appropriate food and clothing purchase decisions.
  5. Housework - doing laundry, washing dishes, dusting, vacuuming, and maintaining a clean place of residence.
  6. Managing medications.
  7. Managing personal finances.
Quality Of Life-AD (QOL-AD) | 8 weeks and 16 weeks
  The QOL-AD is a brief, 13-item measure designed specifically to obtain a rating of the patient's Quality of Life from both the patient and the caregiver. The measure consists of 13 items, rated on a four point scale, with 1 being poor and 4 being excellent. Total scores range from 13 to 52. Items include Memory, Mood, Marriage, Physical Health, etc.
Mini mental state exam (MMSE) | 8 weeks and 16 weeks
  The MMSE is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment.
Falls Efficacy Scale (FES) | 8 weeks and 16 weeks
  On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all, this scale measures how confident the subject is in performing a list of activities without falling.
Activities-specific Balance Confidence Scale (ABC) | 8 weeks and 16 weeks
  Activities-specific balance confidence (ABC) scale is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness. It's a 16-item questionnaire where patients rate their confidence while doing activities. Scoring from 0-100 (0 is no confidence and 100 is full confidence).
Exit-25 | 8 weeks and 16 weeks
  It is a 25-item screening tool that yields a single score reflecting a broad array of executive functions. Each item's possible score ranges from 0 to a maximum of 2 points; total scores range from 0 to 50, with higher scores indicating greater ECF impairment. The items test number/letter sequencing; word and design fluency; sentence-repetition; thematic perception; memory with distraction; interference inhibition; grasp and snout reflexes; social habits; motor perseveration; finger-nose repetition; echopraxia; complex hand sequences; complex commands; counting and serial-order reversal; and automatic, utilization, and imitation behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana P Padala, MD, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebrasaka Medical Center, Omaha, Nebraska, United States